CLINICAL TRIAL: NCT02325765
Title: Corelation Between Circulating Nuclearsome and SIRS Happened After Congential Cardiac Surgery
Brief Title: Study of the Corelation Between Circulating Nuclearsome and SIRS Happened After Congential Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: EY05.055
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Congential Cardiac Surgery
Keywords: congential cardiac surgery; nuclearsome; systemic inflammation response syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Whole Blood, plasma, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- category of RACHS-2 for cardiac surgery: ASD & VSD repair; VSD repair; Tetralogy repair; Tetralogy repair
- category of RACHS-3 for cardiac surgery: DORV repair with or without RV obstruction; AVSD (complete or transitional) repair with or without valve replacement; Coarctation & VSD repair

SUMMARY:
In this study，the investigators want to determine the corelation between circulating nuclearsome and the development of SIRS occured after congenital cardiac surgery, including the serverity of organ damage and inflamation.

DETAILED DESCRIPTION:
Blood was collected from study participants at 6 time points; 1) post-anesthesia induction, 2) post-op hour 0, 3) post-op hour 4, 4) post-op hour 24, 5) post-op hour 48, and 6) post-op hour 72. At each of the 6 time points blood was analyzed for levels of the following:histone,blood routine test , c-reaction protein, procalcitonin, N-terminal pro-brain natriuretic,the hepatorenal function，cardiac function and pulmonary function

ELIGIBILITY:
Inclusion Criteria:

* children with congenial heart disease

Exclusion Criteria:

* Less than 2.5kg
* Prematurity less than 37 weeks estimated gestational age
* Renal failure as described by the pediatric RIFLE criteria

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1-36 months 2.5-15 kilogram accepted congential cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
the perioperation change of histone level | preoperation to 72 hours after congential cardiac surgery

SECONDARY OUTCOMES:
the perioperation change of c-reaction protein level | preoperation to 72 hours after congential cardiac surgery
the perioperation change of cardiac function | preoperation to 72 hours after congential cardiac surgery
the perioperation change of blood routine test | preoperation to 72 hours after congential cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, Study Director — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gao H, Zhang N, Lu F, Yu X, Zhu L, Mo X, Wang W. Circulating histones for predicting prognosis after cardiac surgery: a prospective study. Interact Cardiovasc Thorac Surg. 2016 Nov;23(5):681-687. doi: 10.1093/icvts/ivw198. Epub 2016 Jun 29. PMID 27357468